CLINICAL TRIAL: NCT05203445
Title: Phase II of Neoadjuvant Olaparib in Combination With Pembrolizumab in Patients With Triple Negative Breast Cancer (TNBC) or Hormone Receptor-positive HER2-negative Breast Cancer and Germline Mutations in DNA Damage Repair Genes
Brief Title: A Study of Olaparib and Pembrolizumab in People With Triple Negative Breast Cancer (TNBC) or Hormone Receptor-positive HER2-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-018
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Stage T1c-3N0-3; Olaparib; Pembrolizumab; 21-018
MeSH Terms: conditions — Breast Neoplasms | interventions — olaparib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This trial is designed as a single-arm, open-label, non-randomized study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib in Combination with Pembrolizumab (Experimental): Pembrolizumab 400 mg will be administered as a 30 minute IV infusion every 6 weeks in conjunction with olaparib (for the first 12 weeks) and cytotoxic chemotherapy (after olaparib has been completed) if administered prior to surgery and if the patient is not deemed to have tumor growth.
  Interventions: Drug: Olaparib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Olaparib — Olaparib 300 mg orally BID
Drug: Pembrolizumab — Pembrolizumab 400 mg intravenously q6weeks

SUMMARY:
This study will test any good and bad effects of combining the study drugs pembrolizumab and olaparib, given before the standard surgical procedure, to treat TNBC or HR+ HER2- breast cancers. The study drugs could shrink cancer, but they could also cause side effects. The study researchers want to find out whether the study drugs will shrink the cancer by a certain percentage compared with its current size, which may improve the outcome of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Ability to comply with protocol, in the investigator's judgment
* Newly diagnosed histologically confirmed Stage T1c-3N0-3:

  1. TNBC (ER/PgR negativity will be defined using IHC per ASCO/CAP criteria/HER2-negativity will be defined using ISH or IHC assays per ASCO/CAP criteria) OR
  2. Hormone receptor-positive, HER2-negative breast cancer defined as per ASCO/CAP criteria
* Measurable disease per RECIST v1.1
* Minimum tumor size of 1.5 cm
* All patients must have a germline mutation in BRCA1, BRCA2, PALB2, RAD51C, or RAD51D.
* ECOG Performance Status of 0 or 1
* Patient agreement to undergo appropriate surgical management including, if indicated, axillary lymph node surgery and partial or total mastectomy after completion of neoadjuvant treatment. Note: consideration of neoadjuvant treatment will be determined by disease management team based on the subtypes and minimum size the tumor has to be.
* Baseline LVEF ≥ 53% measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scans
* Have adequate organ function as defined by the following laboratory results obtained within 14 days prior to the first study treatment
* Hematological

  * Absolute neutrophil count (ANC) ≥1500/μL
  * Platelets ≥100 000/μL
  * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
* Renal

  * Creatinine OR ≤1.5 × ULN OR
  * Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* Hepatic

  * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN Patients with known Gilbert syndrome who have serum bilirubin level ≤ 3 X ULN may be enrolled.
  * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) as defined by institutional guidelines OR
  2. A WOCBP who agrees to follow the contraceptive guidance starting at the time of informed consent, during the treatment period and for at least 120 days after the last dose of study treatment (pembrolizumab, olaparib) according to local standard of care.
* Male participants must agree to use contraception starting at the time of informed consent, during the treatment period and for at least 120 days after the last dose of study treatment (pembrolizumab, olaparib) and refrain from donating sperm during this period.

Exclusion Criteria:

* Prior history of invasive breast cancer
* Stage IV (metastatic) breast cancer
* Prior systemic therapy for treatment and prevention of breast cancer
* Contraindication to MRI scan and/or allergy to intravenous contrast-gadolinium
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past X 3 years prior to screening. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical carcinoma in situ are not excluded. Patients with prior ductal/lobular carcinoma in situ are not excluded if they were treated exclusively with mastectomy > 3 years prior to diagnosis of current breast cancer.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab or olaparib and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Severe infections within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment.

  a. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Has a known history of active TB Bacillus Tuberculosis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to study start. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Note: If 72 hours have elapsed between the screening pregnancy test and the performed and must be negative in order for subject to start receiving study medication.
* Patients who have undergone hCG-stimulation for egg harvest as part of fertility preservation within 7 days before treatment initiation are permitted to receive treatment despite a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
pathologically negative MRI-guided biopsy | 12 weeks
  Biopsy-confirmed radiographic complete response will be determined at the 12-week timepoint.
  pCR/RCB0 will be determined at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Gucalp, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm